CLINICAL TRIAL: NCT04607954
Title: MC1923 Phase II Clinical Trial of Durvalumab (MEDI4736) and Lurbinectedin in Patients With Relapsed Extensive Stage Small Cell Lung Cancer Previously Treated With Chemotherapy and Immunotherapy
Brief Title: Durvalumab and Lurbinectedin for the Treatment of Relapsed or Refractory Small Cell Lung Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MC1923; NCI-2020-08088 (Registry Identifier: CTRP (Clinical Trials Reporting Program)); 20-001531 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2020-10-27; First posted 2020-10-29 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Platinum-Resistant Lung Small Cell Carcinoma; Platinum-Sensitive Lung Small Cell Carcinoma; Recurrent Extensive Stage Lung Small Cell Carcinoma; Refractory Extensive Stage Lung Small Cell Carcinoma
MeSH Terms: interventions — durvalumab; Immunoglobulin G; Disulfides; PM 01183

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A (platinum sensitive; progression >3 months) (Experimental): Patients receive durvalumab IV over 60 minutes on day 1 and lurbinectedin IV over 60 minutes on day 1. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Durvalumab; Drug: Lurbinectedin
- Group B (platinum refractory; progression >= 3 months) (Experimental): Patients receive durvalumab IV over 60 minutes on day 1 and lurbinectedin IV over 60 minutes on day 1. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Durvalumab; Drug: Lurbinectedin

INTERVENTIONS:
Biological: Durvalumab — Given IV
  Other Names: Imfinzi; Immunoglobulin G1, Anti-(Human Protein B7-H1) (Human Monoclonal MEDI4736 Heavy Chain), Disulfide with Human Monoclonal MEDI4736 Kappa-chain, Dimer; MEDI-4736; MEDI4736
Drug: Lurbinectedin — Given IV
  Other Names: PM01183; Zepzelca

SUMMARY:
This phase II trial studies the effects of durvalumab and lurbinectedin in treating patients with extensive stage small cell lung cancer that has come back (relapsed) or has not responded to previous treatment with chemotherapy and immunotherapy (refractory). Monoclonal antibodies, such as durvalumab, may interfere with the ability of tumor cells to grow and spread. Lurbinectedin is in a class of medications called alkylating agents. It works by slowing or stopping the growth of cancer cells in the body. Giving durvalumab and lurbinectedin may help kill more tumor cells and help patients live longer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate whether the combination of durvalumab with lurbinectedin can increase the 6-month progression-free survival in patients with extensive stage small cell lung cancer who have progressed after initial combination of chemotherapy and immunotherapy. (Group A and B)

SECONDARY OBJECTIVES:

I. To describe the safety and adverse event profile of each treatment group in patients with extensive stage small cell lung cancer who have progressed after initial combination of chemotherapy and immunotherapy.

II. To assess in a preliminary fashion antitumor efficacy of this approach by assessing overall survival, progression-free survival, and response rate for each treatment group.

CORRELATIVE RESEARCH OBJECTIVE:

I. Blood and tissue will be banked for future studies.

OUTLINE:

Patients receive durvalumab IV over 60 minutes on day 1 and lurbinectedin IV over 60 minutes on day 1. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients without disease progression are followed up at 30 days, every 6 weeks until disease progression, and then every 3 months thereafter for up to 5 years from enrollment. After completion of study treatment, patients with disease progression are followed every 3 months for up to 5 years from enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Histological or cytological confirmation of small cell lung cancer
* Prior treatment requirements:

  * Relapsed or progressed after only one prior chemotherapy and PD-1 or PD-L1 inhibitor regimen
  * Prior therapy must have been an etoposide platinum doublet combined with PD-1 or PD-L1 inhibitor
  * Group 1: Must have "platinum-sensitive" disease according to the following definitions:

    * "Sensitive" disease: Relapse occurred > 90 days after completion of prior therapy
    * "Resistant" Disease: Relapse occurred =< 90 days after completion of prior therapy
  * Group 2: May have "platinum sensitive" (Group 2A) or "platinum resistant" (Group 2B) disease
* Measurable disease
* Body weight > 30 kg
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1
* Hemoglobin >= 9.0 g/dL (obtained =< 15 days prior to registration)
* Absolute neutrophil count (ANC) >= 1500/mm^3 (obtained =< 15 days prior to registration)
* Platelet count >= 100,000/mm^3 (obtained =< 15 days prior to registration)
* Albumin >= 2.5 mg/dL (obtained =< 15 days prior to registration)
* Total bilirubin =< 1.5 x upper limit of normal (ULN) or direct bilirubin =< ULN if total bilirubin is > 1.5 x ULN (obtained =< 15 days prior to registration)
* Alanine aminotransferase (ALT) and aspartate transaminase (AST) =< 2.5 x ULN (=< 5 x ULN for patients with liver involvement) (obtained =< 15 days prior to registration)
* Creatinine OR glomerular filtration rate (GFR) =< 1.5 x ULN OR glomerular filtration rate (GFR) > 60 mL/min for patients with creatinine > 1.5 x ULN (obtained =< 15 days prior to registration)
* Negative pregnancy test done =< 7 days prior to registration, for persons of childbearing potential only
* Persons able to become pregnant OR able to father a child must be willing to use an adequate method of contraception while on treatment and for 120 days after last treatment
* Life expectancy >= 12 weeks
* Provide written informed consent
* Willingness to provide mandatory blood specimens for correlative research
* Willingness to provide mandatory tissue specimens for correlative research
* Willing to return to Mayo Clinic for follow-up (during the active monitoring phase of the study)

Exclusion Criteria:

* Any of the following because this study involves an investigational agent whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown:

  * Pregnant persons
  * Nursing persons
  * Persons of childbearing potential OR able to father a child who are unwilling to employ adequate contraception
* Any of the following prior therapies:

  * Live vaccine < 30 days prior to registration, including intranasal flu vaccine (e.g. Flu-Mist[R]) (Note: Injected seasonal influenza vaccine is not "live")
  * Surgery < 28 days prior to registration
  * Chemotherapy or targeted small molecule therapy < 21 days prior to registration
  * Radiation therapy < 21 days prior to registration
  * Investigational therapy or investigational device < 14 days prior to registration
* Failure to recover to =< grade 1 (or baseline) from adverse events due to previously administered therapies or prior surgery. Exceptions: Neuropathy, fatigue, and/or alopecia may be grade 1
* Known active central nervous system (CNS) metastases. NOTE: Patients with previously treated brain metastases may participate provided all of the following are true:

  * They are stable (without evidence of progression by imaging =< 4 weeks prior to registration and any neurologic symptoms have returned to baseline)
  * Have no evidence of new or enlarging brain metastases, and
  * Are not using steroids =< 14 days prior to registration
* Known leptomeningeal disease
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Known active human immunodeficiency virus (HIV) infection (defined as patients who are not on anti-retroviral treatment and have detectable viral load and CD4+ < 500/ml). NOTE: HIV-positive patients who are well controlled on anti-retroviral therapy are allowed to enroll
* Active autoimmune disease requiring systemic treatment, documented history of severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents. NOTE: Exceptions are allowed for:

  * Vitiligo
  * Resolved childhood asthma/atopy
  * Intermittent use of bronchodilators or inhaled steroids
  * Daily steroids at dose of =< 10mg of prednisone (or equivalent)
  * Local steroid injections
  * Stable hypothyroidism on replacement therapy
  * Stable diabetes mellitus on non-insulin therapy
  * Sjogren's syndrome
* Current or prior use of immunosuppressive medication < 14 days prior to registration. The following are exceptions to this criterion:

  * Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intraarticular injection)
  * Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent
  * Steroids as premedication for hypersensitivity reactions (e.g., premedication for computed tomography [CT] scans)
* Uncontrolled intercurrent illness including, but not limited to:

  * Ongoing or active infection requiring systemic therapy
  * Interstitial lung disease
  * Serious, chronic gastrointestinal conditions associated with diarrhea (e.g., Crohn's disease or others)
  * Known active hepatitis B (i.e., known positive hepatitis B virus [HBV] surface antigen [HBsAg] reactive)
  * Known active hepatitis C (i.e., positive for hepatitis C virus ribonucleic acid [HCV RNA] detected by polymerase chain reaction [PCR])
  * Known active tuberculosis (TB)
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Unstable cardiac arrhythmia or
  * Psychiatric illness/social situations that would limit compliance with study requirements (e.g., substance abuse)
* History of myocardial infarction =< 6 months, or congestive heart failure requiring use of ongoing maintenance therapy for life-threatening ventricular arrhythmias
* Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm
* Hypersensitivity to durvalumab or any of its excipients
* Previous adverse event attributed to durvalumab or other PD-1 or PD-L1 directed therapy that led to drug discontinuation
* History of grade >= 3 immune-related adverse event or any grade of immune-related neurologic or ocular adverse event while receiving immunotherapy. Note: Patients who had endocrine adverse events =< grade 2 are allowed to enroll if they are stable on appropriate replacement therapy and asymptomatic
* Other active malignancy < 6 months prior to registration. EXCEPTIONS: Non-melanotic skin cancer, papillary thyroid cancer, or carcinoma-in-situ of the cervix, or others curatively treated and now considered to be at less than 30% risk of relapse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2020-12-04 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2031-05-01 (Estimated)

PRIMARY OUTCOMES:
6-month progression-free survival rate | At 6 months
  The proportion of successes for 6-month PFS rate will be estimated by the number of successes divided by the total number of evaluable patients. Ninety percent confidence intervals for the true success proportion will be calculated according to the exact binomial method.

SECONDARY OUTCOMES:
Response rate | Up to 5 years
  Proportion of patients with a confirmed tumor response per Response Evaluation Criteria in Solid Tumors (RECIST) and Immune (i)RECIST criteria. Response rate and 90% confidence intervals will be reported or each treatment group separately.
Progression-free survival (PFS) | Up to 5 years
  PFS is defined as the time from registration to the first of either disease progression or death from any cause. Will be estimated using the method of Kaplan-Meier. Medians and 90% confidence intervals will be reported for each treatment group separately.
Overall survival (OS) | Up to 5 years
  OS is defined as the time from registration to death from any cause. Will be estimated using the of Kaplan Meier. Medians and 90% confidence intervals will be reported for each treatment group separately.
Incidence of adverse events (AEs) | Up to 30 days post treatment
  AEs will be monitored using the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. The maximum grade for each type of AE will be recorded for each patient, and frequency tables will be reviewed to determine AE patterns. AEs will be summarized separately for each treatment group.

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos Leventakos, MD, Principal Investigator — Mayo Clinic in Rochester; Anastasios Dimou, MD, Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials